CLINICAL TRIAL: NCT02187094
Title: Study Evaluating the Effect of TC-6499 on Gastric Emptying Time in Diabetic Subjects With Gastroparesis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TC-6499-12-CLP-005
Record Dates: First submitted 2014-06-30; First posted 2014-07-10 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): One capsule of placebo administered as a single dose.
  Interventions: Drug: Placebo
- 2 mg TC-6499 (Experimental): One capsule of 2 mg TC-6499 administered as a single dose.
  Interventions: Drug: TC-6499
- 5 mg TC-6499 (Experimental): One capsule of 5 mg TC-6499 administered as a single dose.
  Interventions: Drug: TC-6499
- 10 mg TC-6499 (Experimental): One capsule of 10 mg TC-6499 administered as a single dose.
  Interventions: Drug: TC-6499

INTERVENTIONS:
Drug: TC-6499
  Arms: 10 mg TC-6499; 2 mg TC-6499; 5 mg TC-6499
Drug: Placebo
  Arms: Placebo

SUMMARY:
Gastroparesis, also referred to as delayed gastric emptying, is a debilitating, chronic disorder that slows or stops the passage of food from the stomach to the small intestine. The purpose of this study is to test whether TC-6499 is safe and effective at reducing gastric emptying time in diabetic subjects with gastroparesis.

DETAILED DESCRIPTION:
This is a 4-way crossover study to assess the effect of TC-6499 on gastric emptying time in diabetic subjects with gastroparesis. The length of study participation for a subject is up to 50 days. During screening, eligible subjects will complete an oral 13-C-spirulina breath test also known as the Gastric Emptying Breath Test (GEBT). During the treatment period, subjects will complete 4 overnight drug assessment visits (treatment arms) where they will receive a randomized single dose of study drug and the GEBT. Each overnight visit will be separated by approximately 7 days. At least 18 subjects will be randomized and complete all 4 dosing arms (actual = 23 randomized subjects and 21 completing all 4 arms of the crossover).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of gastroparesis or symptoms consistent with gastroparesis for at least 6 months (and Gastroparesis Cardinal Symptoms Index total score >22)
* Gastroparesis confirmed using the GEBT
* Type 1 or Type 2 diabetes with a Hemoglobin A1c ≤ 10%
* Fasting blood glucose (finger stick) ≤ 275 mg/dL prior to each GEBT
* Body Mass Index (BMI) ≤ 40
* Willingness to remain in clinical research facility for the protocol-required days of treatment and study procedures
* Willingness to use a double barrier method of birth control (except post-menopausal females)
* Able to understand study procedures and provide written informed consent

Exclusion Criteria:

* History of abdominal surgery including gastric banding procedure
* Chronic parenteral feeding or feeding through a gastrostomy or jejunostomy tube
* Persistent daily vomiting
* A history of eating disorder
* Recent history of poor control of diabetes
* Acute severe gastroenteritis
* Have implanted or use any type of gastric electric stimulator
* Use of opiates, anticholinergic medications, GLP-1 mimetics or amylin analogs
* Use of medications potentially influencing upper gastrointestinal motility or appetite
* Allergies or intolerance to egg, wheat, milk, or algae
* Pregnant or lactating females
* Presence of a clinically significant medical condition at any time during the study
* Presence of clinically significant abnormalities in laboratory findings, physical exam findings or vital signs
* Participated in an investigational drug study within 30 days of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The change in gastric emptying half-time determined for each treatment relative to placebo after single dose administration of study drug in each arm. | 4 hrs post-GEBT meal
  Gastric emptying time will be assessed using the oral 13-C-spirulina breath test also known as the Gastric Emptying Breath Test (GEBT) administered following each treatment.

SECONDARY OUTCOMES:
The percent dose excreted as 13-CO2 at specific post-meal time points for each treatment relative to placebo after single dose administration of study drug in each arm. | 90 and 120 min post-GEBT meal
The time of maximal rate of 13-CO2 expiration for each treatment relative to placebo after single dose administration of study drug in each arm. | 4 hrs post-GEBT meal

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Horizon Research Group, Inc., Mobile, Alabama
  - Prefered Research Partners, Inc., Little Rock, Arkansas
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Ventura Clinical Trials, Ventura, California
  - Wake Research associates, LLC, Raleigh, North Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Aspen Clinical Research, LLC, Orem, Utah